CLINICAL TRIAL: NCT03128931
Title: SedLine Engineering Data Collection Study in Pediatric Patients Undergoing General Anesthesia or Sedation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated as enrollment rate did not meet the requirement of the Sponsor.
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HAMM0001
Record Dates: First submitted 2017-04-14; First posted 2017-04-25 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Group (Experimental): The subjects will be enrolled in the test group and will receive the Pediatric SedLine forehead EEG sensor.
  Interventions: Device: Pediatric SedLine forehead EEG sensor

INTERVENTIONS:
Device: Pediatric SedLine forehead EEG sensor — Pediatric EEG sensor.

SUMMARY:
The purpose of the study is to collect EEG data with the Masimo SedLine device along with vital signs, patient demographics, anesthetic record and surgical procedure during general anesthesia or sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 17 years old and younger
* ASA status I, II, or III.
* Scheduled for surgical and non-surgical procedures scheduled under general anesthesia or sedation (Common procedures include but are not restricted to tonsillectomy, adenoidectomy, urological procedures, dental rehabilitation, orthopedic procedures, biopsies, audiogram, nuclear scans, gastroscopy, colonoscopy, etc. Surgery can be open, laparoscopic, or robotic).

Exclusion Criteria:

* Any deformities or devices that may prevent application of SedLine Array to forehead with a proper fit.
* Cases in which a rapid sequence induction is indicated (emergency, full stomach precautions).
* Subjects who are developmentally delayed.
* Subjects deemed not suitable for study at the discretion of the investigator.

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucille Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: The subjects will be enrolled in the test group and will receive the Pediatric SedLine forehead EEG sensor .
  Pediatric SedLine forehead EEG sensor: Pediatric EEG sensor.
Period: Overall Study
Arm/Group | Test Group
Started | 45
Completed | 41
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Equipment Issues | 3

BASELINE CHARACTERISTICS:
Arm/Group | Test Group
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants For Whom the EEG Data Collection Was Completed
Description: EEG signals will be collected using SedLine sensor for product development under different anesthesia and sedation conditions.
Time Frame: Duration of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group
Number analyzed (Participants) | 41
Participants | 41

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT03128931/Prot_SAP_000.pdf